CLINICAL TRIAL: NCT01493518
Title: A Randomized, Double-blind, Placebo-controlled, Multiple-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Effects of AMG 557 in Subjects With Moderate to Severe Psoriasis
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Effects of AMG 557 in Adults With Psoriasis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20110105
Record Dates: First submitted 2011-08-18; First posted 2011-12-16 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Psoriasis
Keywords: SAFETY; ADULT; PSORIASIS; INFLAMMATION
MeSH Terms: conditions — Psoriasis; Inflammation | interventions — AMG 557

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- PLACEBO (Placebo Comparator)
  Interventions: Drug: AMG 557 or PLACEBO
- AMG 557 (Experimental)
  Interventions: Drug: AMG 557 or PLACEBO

INTERVENTIONS:
Drug: AMG 557 or PLACEBO — Multiple subcutaneous doses of AMG 557 or Placebo on Days 1, 8, 15, 29, 43, 57 and 71.

SUMMARY:
The purpose of this study is to study the safety, tolerability and immunogenicity of AMG 557 following multiple subcutaneous dose administration in adults with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign an Institutional Review Board (IRB)-approved informed consent form (ICF) before any study specific procedures.
* Diagnosis of moderate to severe plaque PsO for at least 6 months prior to screening as defined by:

  * A minimum PASI score of ≥ 10 obtained at screening;
  * Psoriasis involving ≥ 10% of the Body Surface Area (BSA) at screening.
* Received at least 1 previous phototherapy or systemic PsO therapy (but not within the 30 days before study drug administration), or has been a candidate to receive phototherapy or systemic PsO therapy in the opinion of the PI.
* Stable treatment without topical or systemic steroids, topical or systemic retinoids, vitamin D analogues (Dovenex), Psoralen Ultraviolet A (PUVA) therapy, Ultraviolet A (UVA) therapy or Ultraviolet B (UVB) therapy, methotrexate, or cyclosporine for at least 60 days prior to IP administration. Stable treatment of PsO involving scalp, axillae, or groin with topical corticosteroids of moderate strength will be allowed.
* Agrees to wear clothing that protects from sun exposure for the duration of the study.
* Agrees to use sunscreen (SPF of at least 30) on sun-exposed skin for the duration of the study.
* Male or female subjects between 18 and 55 years of age, inclusive at the time of screening.
* Body mass index (BMI) between 18 and 35 kg/m2, inclusive, at screening, unless considered by the PI and the Amgen Medical Monitor to be at an appropriate value in the context of other measured safety parameters.
* Able and willing to complete entire study (including skin biopsies) according to study schedule.
* Additional criteria per protocol.

Exclusion Criteria:

* Diagnosis of guttate, pustular, or other non plaque forms of PsO.
* Evidence of skin conditions other than PsO (eg, eczema) during the screening period that would interfere with evaluations of the effect of IP on PsO.
* Previous receipt of any approved or investigational biologic agent for PsO or other medical conditions.
* Received PUVA therapy, UVA therapy or UVB therapy ≤ 30 days prior to IP administration.
* Treatment with any other systemic PsO therapy or oral or parenteral corticosteroids ≤ 30 days prior to IP administration.
* Use of high potency topical steroids, topical vitamin A or D analog preparations, or anthralin ≤ 30 days prior to IP administration (Note: stable doses > 30 days of low or moderate strength topical steroids are permitted only on the scalp, axillae, and groin according to the package insert).
* Received topical cyclosporin or calcineurin inhibitors such as pimecrolimus (Elidel) and tacrolimus (Protopic) ≤ 30 days prior to IP administration.
* Received IV or oral calcineurin inhibitors such as tacrolimus (Prograf) ≤ 30 days prior to IP administration.
* Significant concurrent medical conditions at the time of screening or prior to randomization, including:

  * Uncontrolled hypertension (defined as screening systolic blood pressure measurement of greater than 140 mm Hg or a screening diastolic blood pressure of greater than 90 mm Hg) confirmed by 2 separate measurements during the screening visit;
  * Unstable angina pectoris;
  * Congestive heart failure;
  * Steroid or oxygen dependent chronic obstructive pulmonary disease;
  * Diagnosis of multiple sclerosis or any other demyelinating disease;
  * Open cutaneous ulcers;
  * Uncontrolled diabetes (HbA1c > 7%).
* History of myocardial infarction.
* Subjects with two or more cardiovascular risk factors (defined as BMI > 30, BP systolic > 140 mm Hg, diagnosis of diabetes, history of cardiovascular event).
* Evidence of significant renal insufficiency during the screening period, defined by a glomerular filtration rate < 50 mL/min using the Cockcroft and Gault equation:

  72 x Serum Creatinine (in mg/dL) / (140 - Age) x Body Weight (in kg) x [0.85 if female]
* Evidence of any bacterial, viral, parasitic, or systemic fungal infections during the 30 days prior to study drug administration (eg, common cold, viral syndrome, flu like symptoms).
* Evidence of a recent (within 6 months of randomization) infection requiring in patient hospitalization or intravenous antibiotics.
* Positive test for HIV antibodies, hepatitis B surface antigen, or hepatitis C antibodies.
* Underlying condition that predisposes the subject to infections (eg, history of splenectomy; history of immunodeficiency).
* Evidence of past or active tuberculosis on chest x-ray performed during screening (or documented evidence on a chest x-ray performed within 6 months prior to planned dosing); known tuberculosis antecedents; known exposure (without adequate treatment) to a person with active tuberculosis; or positive protein purified derivative (PPD) Mantoux skin or serum quantiferon test at screening (without documented history of treatment). A positive result is defined as either induration greater than or equal to 5 mm 48-72 hours after administration (Mantoux) or a positive serum quantiferon test result.
* History of malignancy.
* Evidence of liver disease (eg, serum ALT and AST > 1.5 x the upper limit of normal) during screening period.
* Donated blood (including blood products) or experienced loss of blood ≥ 500 mL within 2 months of screening.
* Additional criteria per protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the number of adverse events per subject, including clinically significant changes in physical examinations, safety lab tests, ECG, vital signs, or immunogenicity to AMG 557 | 28 weeks

SECONDARY OUTCOMES:
Evaluate the efficacy of AMG 557 as measured by the proportion of subjects with a PASI 50, 75 and 90 at week 28 | 28 weeks
Measure the area under the serum concentration curve versus time of AMG 557 after multiple dose administration in subjects with moderate to severe psoriasis | 28 weeks
Measure the peak serum concentration (Cmax) of AMG 557 after multiple dose administration in subjects with moderate to severe psoriasis | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- United States (6):
  - Research Site, Birmingham, Alabama
  - Research Site, Reno, Nevada
  - Research Site, Portland, Oregon
  - Research Site, Dallas, Texas
  - Dallas, Texas
  - Research Site, Salt Lake City, Utah

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com